CLINICAL TRIAL: NCT07150377
Title: A Phase II Single-Arm Study of Iparomlimab and Tuvonralimab (QL1706) in Combination With Lenvatinib and TACE for Advanced Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Shandong First Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-009
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvonralimab in combination with Lenvatinib and TACE for advanced hepatocellular car (Experimental)
  Interventions: Drug: First-line Cohort; Drug: Second-line Cohort

INTERVENTIONS:
Drug: First-line Cohort — Iparomlimab and Tuvonralimab: 7.5 mg/kg, IV, Q3W Lenvatinib: 12 mg (for body weight ≥60 kg) or 8 mg (for body weight ≤60 kg), po, qd
Drug: Second-line Cohort — Iparomlimab and Tuvonralimab: 7.5 mg/kg, IV, Q3W Lenvatinib: 12 mg (for body weight ≥60 kg) or 8 mg (for body weight ≤60 kg), po, qd

SUMMARY:
To evaluate the efficacy of Iparomlimab and Tuvonralimab in combination with Lenvatinib and TACE for advanced hepatocellular carcinoma by assessing Progression-Free Survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* First-line Cohort:

  1. Confirmed diagnosis of hepatocellular carcinoma (HCC), aged > 18 years. No prior systemic therapy.
  2. Child-Pugh class A/B at baseline.
  3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment.
  4. Measurable lesions per modified Response Evaluation Criteria in Solid Tumors (mRECIST).
  5. Adequate organ and bone marrow function.

Second-line Cohort:

1. Confirmed diagnosis of HCC, aged > 18 years.
2. Prior first-line therapy (including targeted therapy or immunotherapy).
3. Child-Pugh class A/B at baseline.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment.
5. Measurable lesions per modified Response Evaluation Criteria in Solid Tumors (mRECIST).
6. Adequate organ and bone marrow function.

Exclusion Criteria:

1. Concomitant hepatic encephalopathy.
2. History of any nephrotic syndrome.
3. History of clinically significant cardiovascular disease or arterial thromboembolic events, including stroke, myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack within 6 months prior to randomization.
4. Evidence of any prior or current coagulopathy or bleeding diathesis, or any type of surgery performed within the past 28 days (biopsy is not excluded).
5. History of abdominal fistula, gastrointestinal perforation, refractory non-healing gastric ulcer, or active gastrointestinal bleeding within 6 months prior to randomization.
6. Main portal vein thrombosis visible on baseline imaging.
7. Pleural or peritoneal effusion requiring clinical intervention.
8. Gastroesophageal varices.
9. Portal vein invasion (VP3 or VP4).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-08-24 (Estimated); Primary Completion 2026-08-24 (Estimated); Study Completion 2028-08-24 (Estimated)

PRIMARY OUTCOMES:
PFS | 1 year
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse

SECONDARY OUTCOMES:
OS | 2 years
  Time from randomization to death from any cause
Objective Response Rate | 1 year
  It refers to the proportion of patients (mainly solid tumors) whose tumor has shrunk to a certain extent and remained there for a certain period of time, including Complete Response (CR) and Partial Response (PR)
Adverse Events | 2 years
  It refers to all adverse medical events that occur after a subject receives an investigational drug, which may be manifested as symptoms, signs, diseases, or abnormalities in laboratory tests, but may not necessarily be causally related to the investigational drug It refers to all adverse medical events that occur after a subject receives an investigational drug, which may be manifested as symptoms, signs, diseases, or abnormalities in laboratory tests, but may not necessarily be causally related to the investigational drug It refers to all adverse medical events that occur after a subject receives an investigational drug, which may be manifested as symptoms, signs, diseases, or abnormalities in laboratory tests, but may not necessarily be causally related to the investigational drug

CONTACTS AND LOCATIONS:
Overall Officials: yan hai Liu, Principal Investigator — The Second Affiliated Hospital of Shandong First Medical University

IPD SHARING:
Plan to Share IPD: No